CLINICAL TRIAL: NCT03995680
Title: Efficacy and Safety of a New Chewable Tablet of Mebendazole Versus the Swallowable, Standard Tablet of Mebendazole Against Hookworm Infections in Children: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of a New Chewable Versus the Swallowable Tablet of Mebendazole Against Hookworm
Acronym: CHEW_MEB_PEMBA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Public Health Laboratory Ivo de Carneri (Other)
Responsible Party: Principal Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEW_MEB
Record Dates: First submitted 2019-05-30; First posted 2019-06-24 (Actual); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Hookworm Infections
Keywords: Mebendazole; Chewable tablet; Hookworm; Soil-transmitted helminths; Efficacy; Safety; Acceptability
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis | interventions — Mebendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Chewable tablet of mebendazole (Experimental): * 3-5 year olds allocated to the swallowable tablet arm will be given the crushed tablet on a spoon mixed with a small amount of clean water;
  * 6-12 year olds allocated to the swallowable tablet arm will be given the whole tablet to swallow with a glass of clean water;
  Interventions: Drug: Mebendazole
- Swallowable tablet of mebendazole (Active Comparator): * 3-5 year olds allocated to the chewable tablet arm will be encouraged to chew the tablet and swallow it without water; if they cannot chew it then a small amount of water will be added to the tablet in a spoon;
  * 6-12 year olds allocated to the chewable tablet arm will be encouraged to chew the tablet and then swallow it without water.
  Interventions: Drug: Mebendazole

INTERVENTIONS:
Drug: Mebendazole — Treatment with one of the two formulations of mebendazole. The only difference between both arms is the type of formulation of the drug: chewable versus swallowable tablet.

SUMMARY:
The rational of this study is to provide evidence on the safety and efficacy of a new chewable tablet of mebendazole compared to the standard tablet in preschool- and school-aged children infected with hookworm.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children aged between 3 and 12 years;
* Written informed consent signed by caregiver;
* Was examined by a study physician before treatment;
* Provided two stool samples at baseline;
* Hookworm EPG > 100 and at least two Kato-Katz thick smears slides with more than one hookworm egg;

Exclusion Criteria:

* Pregnant;
* Presence or history of major systemic or chronic illnesses, as assessed by a medical doctor, such as can upon initial clinical assessment;
* Suffers from severe anemia (Hb < 80 g/l);
* Received anthelminthic treatment or metronidazole within past four weeks.
* Attending other clinical trials during the study.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 397 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keiser, PhD, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (1):
- Public Health Laboratory Ivo de Carneri, Chake Chake, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmeirim MS, Bosch F, Ame SM, Ali SM, Hattendorf J, Keiser J. Efficacy, safety and acceptability of a new chewable formulation versus the solid tablet of mebendazole against hookworm infections in children: An open-label, randomized controlled trial. EClinicalMedicine. 2020 Sep 20;27:100556. doi: 10.1016/j.eclinm.2020.100556. eCollection 2020 Oct. PMID 33150325

RESULTS

PARTICIPANT FLOW:
Groups:
- Chewable Tablet of Mebendazole: A single 500 mg dose of the new chewable mebendazole tablets will be administered to each child in this arm.
  Mebendazole: Treatment with one of the two formulations of mebendazole. The only difference between both arms is the type of formulation of the drug: chewable versus swallowable tablet.
- Swallowable Tablet of Mebendazole: A single 500 mg dose of the standard swallowable mebendazole tablets will be administered to each child in this arm.
  Mebendazole: Treatment with one of the two formulations of mebendazole. The only difference between both arms is the type of formulation of the drug: chewable versus swallowable tablet.
Period: Overall Study
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
Started | 199 | 198
Completed | 197 | 196
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole | Total
Number analyzed (Participants) | 197 | 196 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (2.0) | 9.4 (2.1) | 9.3 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 80 | 167
  Male | 110 | 116 | 226
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: centimeters] | 130.5 (11.5) | 130.8 (11.6) | 130.7 (11.6)
Weight [Mean (Standard Deviation); unit: kilograms] | 25.4 (6.3) | 26.0 (6.6) | 25.7 (6.5)
Hemoglobin [Mean (Standard Deviation); unit: grams per liter] | 121.5 (10.3) | 123.5 (10.7) | 122.5 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Egg Reduction Rate (ERR) of the Two Formulations of Mebendazole Against Hookworm
Description: Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. The egg reduction rate (ERR) is calculated as follows: ERR = (1-(geometric mean EPG at follow-up/geometric mean EPG at baseline))*100). Note: in contrast to the publication the "outcome measure" entry mask requires the complementary percentage: (geometric mean at follow-up/geometric mean at baseline)*100).
Time Frame: Baseline (before treatment) and sometime between 14 and 21 days post-treatment
Measure: Number (95% Confidence Interval); unit: percentage change in hookworm egg counts
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
Number analyzed (Participants) | 197 | 198
percentage change in hookworm egg counts | 68.5 [60.4 to 75.3] | 70.8 [63.5 to 76.7]

2. Secondary Outcome: Cure Rate (CR) of Mebendazole Against Hookworm
Description: Cure rates (CRs) will be calculated as the percentage of egg-positive participants at baseline who become egg-negative after treatment.
Time Frame: Baseline (before treatment) and sometime between 14 and 21 days post-treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
Number analyzed (Participants) | 197 | 196
percentage of participants | 12.7 [8.4 to 18.2] | 11.2 [7.2 to 16.5]

3. Secondary Outcome: CR of Both Mebendazole Regimens Against Trichuris Trichiura
Description: as for outcome 2
Time Frame: Baseline (before treatment) and sometime between 14 and 21 days post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
Number analyzed (Participants) | 197 | 196
percentage of participants | 9.8 | 7.3

4. Secondary Outcome: Geometric ERR of Both Mebendazole Formulations Against Trichuris Trichiura
Description: as for outcome 1
Time Frame: Baseline (before treatment) and sometime between 14 and 21 days post-treatment
Measure: Number (95% Confidence Interval); unit: percentage change in T. trich egg counts
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
Number analyzed (Participants) | 197 | 196
percentage change in T. trich egg counts | 73.3 [65.7 to 79.4] | 74.2 [67.2 to 79.8]

5. Secondary Outcome: CR of Both Mebendazole Formulations Against Ascaris Lumbricoides
Description: as for outcome 2
Time Frame: Baseline (before treatment) and sometime between 14 and 21 days post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
Number analyzed (Participants) | 197 | 196
percentage of participants | 95.3 | 97.8

6. Secondary Outcome: Geometric ERR of Both Mebendazole Formulations Against Ascaris Lumbricoides.
Description: as for outcome 1
Time Frame: Baseline (before treatment) and sometime between 14 and 21 days post-treatment
Measure: Number; unit: percentage change in A. lumbr egg counts
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
Number analyzed (Participants) | 197 | 196
percentage change in A. lumbr egg counts | 99.9 | 99.9

7. Secondary Outcome: Arithmetic ERR of the Two Formulations of Mebendazole Against Hookworm
Description: Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. The egg reduction rate (ERR) is calculated as follows: ERR = (1-(arithmetic mean EPG at follow-up/arithmetic mean EPG at baseline))*100). Note: in contrast to the publication the "outcome measure" entry mask requires the complementary percentage: (arithmetic mean at follow-up/arithmetic mean at baseline)*100).
Time Frame: Baseline (before treatment) and sometime between 14 and 21 days post-treatment
Measure: Number (95% Confidence Interval); unit: percentage change in hookworm egg counts
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
Number analyzed (Participants) | 197 | 196
percentage change in hookworm egg counts | 38.2 [26.6 to 47.8] | 28.1 [8.5 to 44.3]

8. Secondary Outcome: Arithmetic ERR of Both Mebendazole Formulations Against Trichuris Trichiura
Description: as for outcome 7
Time Frame: Baseline (before treatment) and sometime between 14 and 21 days post-treatment
Measure: Number; unit: percentage change in T. trich egg counts
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
Number analyzed (Participants) | 197 | 196
percentage change in T. trich egg counts | 52.9 | 50.9

9. Secondary Outcome: Arithmetic ERR of Both Mebendazole Formulations Against Ascaris Lumbricoides
Description: as for outcome 7
Time Frame: Baseline (before treatment) and sometime between 14 and 21 days post-treatment
Measure: Number; unit: percentage change in A. lumbr egg counts
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
Number analyzed (Participants) | 197 | 196
percentage change in A. lumbr egg counts | 98.7 | 99.8
Statistical Analysis 1: Comparison: Chewable Tablet of Mebendazole vs Swallowable Tablet of Mebendazole; The 95% confidence intervals (CIs) for ERRs and the difference between ERRs were estimated via bootstrap resampling. Superiority was claimed if the 95% confidence interval of the difference in ERRs did not include unity. Logistic regression models were used to assess efficacy in terms of CRs. In a subsequent analysis an adjusted logistic regression (adjustment for age, sex, weight and baseline infection intensity) was performed; Test type: Superiority; Regression, Logistic; Adjusted for age, sex, weight and baseline hookworm infection intensity (light or moderate/heavy); Difference in Egg Reduction Rate (%) = 2.3, 95% CI 2-sided [-7.8 to 12.6]

ADVERSE EVENTS:
Time Frame: 3 hours and 24 hours post-treatment
Description: Physicians and nurses actively questioned each child for adverse events using a questionnaire
Arm/Group | Chewable Tablet of Mebendazole | Swallowable Tablet of Mebendazole
All-Cause Mortality (participants affected / at risk) | 0/197 | 0/196
Serious Adverse Events (participants affected / at risk) | 0/197 | 0/196
Other Adverse Events (participants affected / at risk) | 14/197 | 15/196
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chewable Tablet of Mebendazole (N=197) | Swallowable Tablet of Mebendazole (N=196)
Abdominal pain (General disorders) | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03995680/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT03995680/ICF_001.pdf